CLINICAL TRIAL: NCT03319056
Title: Cardiopulmonary Health Effects of Indoor Air Purification and Different Indoor Environmental Factors Among School Children in Beijing
Brief Title: Indoor Air and Children Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Furong Deng, MD & PhD, Professor, Deputy Director of Department of Occupational & Environmental Health Sciences, Peking University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FDeng17
Record Dates: First submitted 2017-10-18; First posted 2017-10-24 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Cardiopulmonary Disease
MeSH Terms: conditions — Pulmonary Heart Disease | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real purification (Active Comparator): Air purifier turned on
  Interventions: Other: Air purifier
- Sham purification (Sham Comparator): Air purifier turned off
  Interventions: Other: Air purifier

INTERVENTIONS:
Other: Air purifier — active- or sham-mode air purifier used in 6 classrooms in a school with a crossover design

SUMMARY:
The objective of this study is to investigate the cardiopulmonary health effects of indoor air purification and different indoor environmental factors among school students in Beijing.

DETAILED DESCRIPTION:
This randomized, double-blind crossover study was conducted to explore the cardiopulmonary effects of ionization air purification among 48 children in Beijing. Real or sham purification was performed in classrooms for 5 weekdays in a random order with a 2-month wash-out period. During the study periods, different indoor environmental factors were monitored including size-fractionated particulate matter (PM), black carbon (BC), ozone, carbon dioxide (CO2), negative air ions (NAI), noise, temperature and relative humidity, which were controlled as confounders in the analysis of the effects of indoor air purification. In addition, we analyzed the cardiopulmonary effects of those environmental factors on the children.

ELIGIBILITY:
Inclusion Criteria:

* living in Beijing for more than two consecutive years;
* living in school dormitories from Monday to Friday.

Exclusion Criteria:

* suffering any health condition;
* having asthma or thoracic surgery history.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Levels of lung function indicators | 10 weekdays for intervention (active or sham) and 2 wash-out months
  Lung function test was conducted including forced expiratory volume in one second (FEV1) and peak expiratory flow (PEF).

SECONDARY OUTCOMES:
Changes in autonomic cardiac function | 10 weekdays for intervention (active or sham) and 2 wash-out months
  Ambulatory electrocardiogram (ECG) was monitored including heart rate (HR) and heart rate variability (HRV).
Level of respiratory inflammation | 10 weekdays for intervention (active or sham) and 2 wash-out months
  Fractional exhaled nitric oxide (FeNO) test was conducted.
Changes in ST-segment elevation | 10 weekdays for intervention (active or sham) and 2 wash-out months
  Ambulatory electrocardiogram (ECG) was monitored.
Levels of oxidative stress in Exhaled Breath Condensate (EBC) | 10 weekdays for intervention (active or sham) and 2 wash-out months
  EBC was collected using a designated device for oxidative stress analysis.
Levels of urinary metabolomics | 10 weekdays for intervention (active or sham) and 2 wash-out months
  Urine samples were collected for metabolomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Furong Deng, PhD&MD, Principal Investigator — Peking University
Locations (1):
- School of Pubic Health, Peking University, Beijing, Beijing Municipality, China